CLINICAL TRIAL: NCT06996106
Title: Effect of Platelet Rich Fibrin on Septoplasty :A Comparative Study
Brief Title: Outcomes of PRF on Septoplasty in Patient With Nasal Septal Deviation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Ibrahim Abdallah Abdel wahd Abo Hussein, ahmed ibrahim, Kafrelsheikh University
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PRF in septoplasty
Record Dates: First submitted 2025-05-02; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Nasal Septum; Deviation; Nasal Septal Srur

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- platelet rich fibrin (Active Comparator): usage of platelet rich fibrin in this arm underging setoplasty
  Interventions: Other: Effect of Platelet Rich Fibrin on Septoplasty
- control group (Active Comparator): traditional septoplasty
  Interventions: Other: Effect of Platelet Rich Fibrin on Septoplasty

INTERVENTIONS:
Other: Effect of Platelet Rich Fibrin on Septoplasty — it is a randomized trial of usage of platelet rich fibrin in septoplasty

SUMMARY:
The aim of this study is to assess the effectiveness of Platelet-Rich Fibrin (PRF) in improving postoperative healing, reducing complications, and enhancing functional outcomes in patients undergoing septoplasty

DETAILED DESCRIPTION:
Septoplasty is a routine surgical intervention to correct nasal septal deviation, a major cause of nasal obstruction and chronic sinusitis. Despite advancements, postoperative complications-such as mucosal injury, synechiae, septal perforation, and hematoma-continue to impact outcomes and patient satisfaction.

Platelet-rich fibrin (PRF), first described by Choukroun et al., represents an autologous biomaterial rich in growth factors like PDGF, TGF-β, VEGF, and IGF-1, known to accelerate wound healing and tissue regeneration. Unlike platelet-rich plasma (PRP), PRF is easier to prepare, does not require anticoagulants, and forms a fibrin matrix conducive to sustained release of cytokines.

Several studies across disciplines-oral surgery, dermatology, orthopedics-support the regenerative potential of PRF. In nasal surgery, the delicate mucosal environment could benefit significantly from enhanced healing facilitated by PRF.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years undergoing septoplasty. Presence of cartilage deviated nasal septum requiring repair. No contraindications to PRF therapy.

Exclusion Criteria:

* History of coagulopathy or anticoagulant therapy. Active infection or systemic disease. Known hypersensitivity to PRF components. Previous nasal surgery Autoimmune or systemic inflammatory disease

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Effect of submucoperichondrial application of platelet rich fibrin on healing of nasal septum mucosa after septoplasty | postoperative at 1st week , 1st month , 3rd month
  Mucosal Healing will be assessed by visual nasal endscope

IPD SHARING:
Plan to Share IPD: No